CLINICAL TRIAL: NCT07391670
Title: A Phase I, Multicentre, Dose Escalation and Dose Expansion Study to Investigate the Pharmacokinetics and Safety of Subcutaneous Durvalumab in Adult Participants With Solid Tumours
Brief Title: A Phase I Dose Escalation and Dose Expansion Study to Investigate the Pharmacokinetics and Safety of Subcutaneous Durvalumab
Acronym: IMFINZI-subQ
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D907HC00001; 2025-521639-34-00 (Other: EU CT number)
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumours
Keywords: Pharmacokinetics; Non-small cell lung cancer (Stage III, unresectable); Small cell lung cancer (Limited stage); Hepatocellular carcinoma (Unresectable); Subcutaneous; Human hyaluronidase; Monoclonal antibody; Programmed cell death ligand 1 (PD-L1); Programmed cell death protein 1; Anticancer therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Carcinoma, Hepatocellular | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: SC Durvalumab DL1 (Experimental): Participants will receive DL1 of SC durvalumab + rHu followed by IV durvalumab at predefined intervals.
  Interventions: Drug: SC durvalumab + rHu; Drug: IV durvalumab; Drug: Tremelimumab
- Part 1: SC Durvalumab DL2 (Experimental): Participants will receive DL2 of SC durvalumab + rHu followed by IV durvalumab at predefined intervals.
  Interventions: Drug: SC durvalumab + rHu; Drug: IV durvalumab; Drug: Tremelimumab
- Part 2: Expansion Cohort, SC Durvalumab Dose Level X (Experimental): Participants will receive dose level X (determined from data analysis in Part 1) of SC durvalumab + rHu followed by IV durvalumab at predefined intervals.
  Interventions: Drug: SC durvalumab + rHu; Drug: IV durvalumab; Drug: Tremelimumab

INTERVENTIONS:
Drug: SC durvalumab + rHu — Durvalumab + rHu will be administered subcutaneously.
Drug: IV durvalumab — Durvalumab will be administered intravenously.
  Other Names: MEDI4736
Drug: Tremelimumab — Tremelimumab will be administered to participants with unresectable HCC as an IV infusion.

SUMMARY:
The purpose of the study is to determine a subcutaneous (SC: under the skin) durvalumab + recombinant human hyaluronidase (rHu) dose that yields systemic drug exposure similar to intravenous (IV: into the veins) durvalumab administration and to evaluate the pharmacokinetics and safety of SC durvalumab + rHu injection in participants with different types of solid tumours (cancers).

DETAILED DESCRIPTION:
This is a Phase I, multicentre study that will consist of 2 parts -

* Part 1: Dose Escalation
* Part 2: Dose Expansion

Part 1 may include participants with solid tumours - non-small cell lung cancer (NSCLC), hepatocellular carcinoma (HCC) or limited-stage small cell lung cancer (LS-SCLC). It will further consist of 2 planned dose levels of SC durvalumab - Dose level 1 (DL1) and Dose level 2 (DL2).

Part 2 will include participants with unresectable HCC. It will be initiated once a dose has been identified based on Part 1.

ELIGIBILITY:
Inclusion Criteria:

* An Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy of ≥ 12 weeks at enrolment.
* Adequate organ and marrow function.
* Minimum body weight > 30 kg.

Part 1 only:

Locally Advanced Unresectable (Stage III) NSCLC Participants -

* Histological or cytological documented evidence of NSCLC (locally advanced, unresectable, Stage III).
* Must have received at least 2 cycles of platinum-based chemotherapy concurrent with definitive radiation therapy.
* Have not progressed following definitive concurrent chemoradiation.

LS-SCLC Participants -

* Histologically or cytologically documented LS-SCLC (Stage I-III).
* Received 4 cycles of chemotherapy concurrent with radiotherapy, which must be completed within 1 to 42 days prior to enrolment.
* Have not progressed following definitive concurrent chemoradiation.

Part 1 and 2:

Unresectable HCC Participants -

* Unresectable HCC based on histopathological confirmation.
* No prior systemic therapy for unresectable HCC.
* Must not be eligible for locoregional therapy for unresectable HCC.
* Child-Pugh Score class A.
* Measurable disease as defined by RECIST v1.1.

Exclusion Criteria:

* Active or prior documented autoimmune disease requiring systemic treatment.
* Uncontrolled infection (including human immunodeficiency virus [HIV], hepatitis B or C).
* Prior exposure to immune checkpoint inhibitors.

Part 1 only:

Locally Advanced Unresectable (Stage III) NSCLC Participants -

* Mixed SCLC and NSCLC histology.
* Active pneumonitis or interstitial lung disease requiring systemic therapy.

LS SCLC Participants -

* Mixed SCLC and NSCLC histology.
* Extensive-stage disease.
* History of Grade ≥ 2 pneumonitis.

Part 1 and 2:

Unresectable HCC Participants -

* Hepatic encephalopathy.
* Uncontrolled ascites.
* Active gastrointestinal (GI) bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration-time curve | From first dose of study intervention (Day 1), at predefined intervals throughout the administration of durvalumab (approximately 17 months).
  To characterise the AUC of SC durvalumab.
Observed lowest concentration before the next dose is administered (Ctrough) | From first dose of study intervention (Day 1), at predefined intervals throughout the administration of durvalumab (approximately 17 months).
  To characterise the Ctrough of SC durvalumab

SECONDARY OUTCOMES:
Area under the concentration-time curve from time 0 to last quantifiable concentration (AUClast) | From first dose of study intervention (Day 1), at predefined intervals throughout the administration of durvalumab (approximately 17 months).
  To characterise the AUClast of SC durvalumab.
Maximum observed concentration (Cmax) | From first dose of study intervention (Day 1), at predefined intervals throughout the administration of durvalumab (approximately 17 months).
  To characterise the Cmax of SC durvalumab.
Time to reach maximum concentration following drug administration (tmax) | From first dose of study intervention (Day 1), at predefined intervals throughout the administration of durvalumab (approximately 17 months).
  To characterise the tmax of SC durvalumab.
Terminal elimination half-life (t1/2λz) | From first dose of study intervention (Day 1), at predefined intervals throughout the administration of durvalumab (approximately 17 months).
  To characterise the t1/2λz of SC durvalumab.
Total body clearance/apparent total body clearance (CL[/F]) | From first dose of study intervention (Day 1), at predefined intervals throughout the administration of durvalumab (approximately 17 months).
  To characterise the CL(/F) of SC durvalumab.
Apparent volume of distribution based on the terminal phase volume (Vz[/F]) | From first dose of study intervention (Day 1), at predefined intervals throughout the administration of durvalumab (approximately 17 months).
  To characterise the VZ(/F) of SC durvalumab.
Average drug concentration over a dosing interval (Cavg) | From first dose of study intervention (Day 1), at predefined intervals throughout the administration of durvalumab (approximately 17 months).
  To characterise the Cavg of SC durvalumab.
Serum concentration of durvalumab | From first dose of study intervention (Day 1), at predefined intervals throughout the administration of durvalumab (approximately 17 months).
  To characterise the serum concentration of SC durvalumab at specified timepoints.
Number of participants with adverse events (AEs) | Up to Survival Follow-up (approximately 17 months)
  To assess the safety and tolerability of SC durvalumab.
Number of participants with dose-limiting toxicities (DLTs) | Up to Survival Follow-up (approximately 17 months)
  To assess the safety and tolerability of SC durvalumab.

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/